CLINICAL TRIAL: NCT01372930
Title: The Safety and Efficacy of Etanercept in Treating Patient With Acute ST Segment Elevated Myocardial Infarction
Brief Title: Etanercept Treating Patient With Acute ST Segment Elevated Myocardial Infarction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Ling Tao, Department of Cardiology of Xijing Hospital; Fourth Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: xjyy110504
Record Dates: First submitted 2011-06-10; First posted 2011-06-14 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2010-03

CONDITIONS: Myocardial Infarction
Keywords: Etanercept; acute ST segment elevated myocardial infarction; percutaneous coronary intervention; myocardial reperfusion injury
MeSH Terms: conditions — Myocardial Infarction; Myocardial Reperfusion Injury | interventions — Etanercept; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etanercept (Experimental)
  Interventions: Drug: Etanercept
- saline (Placebo Comparator)
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Etanercept — Etanercept 25mg in 1ml(subcutaneous injection)at 2h and 72h after PCI
  Other Names: Enbrel
  Arms: Etanercept
Drug: saline — saline 1ml(subcutaneous injection) at 2h and 72h after PCI
  Arms: saline

SUMMARY:
Our aim is to observe whether anti-TNF-alpha regimen will effect serum adiponectin concentration after myocardial infarction/reperfusion and also beneficial for the patients undergoing percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Ischemic/reperfusion injury in patients with acute myocardial infarction (AMI) undergoing percutaneous coronary intervention (PCI) is associated with increased inflammatory cytokines that including TNF-alpha that can exert deleterious effects and therefore contribute to cardiac dysfunction and cardiomyocytes apoptosis. Several studies on rodents have reported administration of sTNFR-Fc, a scavenger of the pro-inflammatory cytokine TNF-alpha at the time of reperfusion would protect against ischemic/reperfusion injury. Also reports had shown that serum TNF-alpha concentration is negatively correlated with a cardioprotective cytokine adiponectin. Adiponectin (Ad) is an abundant protein hormone regulatory of numerous metabolic processes. The major intracellular pathway activated by Ad includes phosphorylation of AMP-activated protein kinase, which is responsible for many of Ad's metabolic regulatory, anti-inflammatory, vascular protective, and anti-ischemic properties. The aim of the present study was to verify whether the administration of Etanercept, an FDA approved rheumatoid arthritis treating sTNFR-Fc, at the reperfusion time would protect against ischemic/reperfusion injury on patient, and effect serum adiponectin level.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute ST segment elevated myocardial infarction in 12h

Exclusion Criteria:

* Cardiogenic shock
* old myocardial infarction
* other causes of cardiac insufficiency
* tumor
* Coronary anatomy unsuitable for PCI or Need of emergency coronary artery by-pass grafting
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-04; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Composite of major adverse cardiovascular events (MACE) consisting of cardiovascular death, fatal myocardial infarction and fatal stroke | 30 days

SECONDARY OUTCOMES:
Composite endpoint of major cardiovascular events, non-elective coronary revascularization procedures and hospitalization for unstable angina Cardiovascular death Non-fatal myocardial infarction Non-fatal stroke of all classifications | 30 days
Elevation of ALT, AST and CK | 30 days
serum adiponectin concentration, activity and isoforms | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China